CLINICAL TRIAL: NCT01597024
Title: Full4Health: Neuro-gut Interactions in Humans Across the Lifecourse
Brief Title: Full4Health: Understanding Food-gut-brain Axis Across the Lifecourse
Acronym: F4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Daniel Crabtree, Research Fellow, University of Aberdeen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Full4Health
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Obesity
Keywords: appetite; food; gut; brain; satiety; hunger; gut hormones
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1: Breakfast Study (Experimental)
  Interventions: Other: Breakfast Study
- Phase 2: fMRI Study (Experimental)
  Interventions: Other: fMRI Study

INTERVENTIONS:
Other: Breakfast Study — Participants (male and female, lean and obese, children, teenagers, adults, and elderly) will take part in 4 morning sessions, consuming a test breakfast milk based beverage and appetite. Biomarkers in blood will be measured and behavioural questionnaires completed. We will also collect a single saliva sample from each participant to examine genetic traits related to appetite, food choice, body weight, and energy expenditure. There will be two milk based beverages, one protein enriched (30% protein from calories) and one normal protein (15% protein). Participants will be offered a morning snack buffet to assess ad libitum energy intake. Phase 1 will also include a subgroup of malnourished male and female elderly participants. However, this group will only complete two morning sessions during which they will consume a low protein and a high protein milk based beverage. Appetite will be recorded and libitum energy intake will be measured. In addition, 24hr energy intake will be recorded.
  Arms: Phase 1: Breakfast Study
Other: fMRI Study — We will fMRI scan normal weight and overweight subjects of both gender from the four different age groups only: 8-10, 13-17, 24-45 and 65-75 years. Participants will be measured twice, on separate days, either after an overnight fast or after a test meal, fed to satiation (because hunger will modulate the response to food presentation). The participants will conduct a computerised task that will be performed in the scanner to assess hedonic responses to food cues. Physiological biomarkers will be measured during both trials for the assessment of appetite hormone circulation. Saliva samples will be taken for DNA analysis. DNA extraction techniques will be used to examine genetic traits linked to appetite, food choice, body weight, and energy expenditure.
  Arms: Phase 2: fMRI Study

SUMMARY:
The primary aim of this work is, to 'relate psychological and behavioural parameters of hunger/satiety and food preference to gut hormones, neural activation and energy metabolism by dietary manipulation, across the human lifespan'.

DETAILED DESCRIPTION:
The Full4Health project aims to further understanding of the mechanisms of hunger and satiety. The proposal integrates investigation of human volunteers and laboratory rodents throughout the life course, applying imaging and other cutting edge technologies to critical research questions. Full4Health will combine study of the mechanisms of hunger and satiety with intervention studies to validate the effects of the relevant food characteristics on the regulation of satiety/hunger. The development of cerebral responses to food through the gut-brain axis across lifespan particularly during childhood, adolescence and elderly will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the fMRI study
* Right-handed
* Not heavy smokers (less 10 day)
* MRI compatibility:
* no claustrophobia
* no metal in the body (including dental braces)

Exclusion Criteria:

* Heavy smokers (more than 10/day)
* Morbid obese (BMI>40 kg/m2)
* Pregnancy
* Obesity of known endocrine origin
* Neurological disorders including Cerebral Palsy
* Alzheimers disease
* Multiple Sclerosis
* Parkinsons disease
* Medication known to influence appetite (orlistat, oral antidiabetics, insulin, digoxin, anti-arrhythmics, sibutramine, antidepressants)
* Self report fever/systemic infection
* Inability to participate in fMRI scanning sessions including contraindications to MRI
* Participation in medical or surgical weight loss programme within 1 month of selection
* History of cerebrovascular disease
* Current major depressive disorder, bipolar disorder or past history of suicide attempt or self harm
* History of drug or alcohol misuse
* History of significant cardiovascular disease
* Allergy to any of the breakfasts components.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in concentrations of biomarkers of appetite in response to each milk-based beverage | During each of the four 'Breakfast Study' visits blood will be taken at baseline, and 30, 60, and 120 minutes after consuming the milk-based beverage. Each visit will be seperated by one week.
  The following blood-borne biomarkers of appetite will be measured:
  * Glucose
  * Total cholesterol
  * Triglycerides
  * Low density lipoprotein
  * High density lipoprotein
  * Insulin
  * Ghrelin (active)
  * Glucagon-like peptide-1 (active)
  * Peptide YY (total)
  * Leptin

SECONDARY OUTCOMES:
Neural responses to images of food when fasted and after consuming a milk-based beverage | There will be one week between both conditions (fasted and fed)
  The subjects will conduct a computerised task that will be performed in the functional magnetic resonance imaging (fMRI) scanner. Subjects will be measured twice, on separate days, either after an overnight fast or after a test meal fed to satiation.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, PhD, Principal Investigator — The Rowett Institute of Nutrition and Health, University of Aberdeen
Locations (3):
- Harokopia Univeristy, Athens, Greece
- University Medical Center Utrecht, Utrecht, Netherlands
- The Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, Aberdeenshire, United Kingdom

REFERENCES:
- [Derived] Crabtree DR, Buosi W, Fyfe CL, Horgan GW, Holst JJ, Johnstone AM; Full4Health-study Group. Salivary ghrelin response to drinks varying in protein content and quantity and association with energy intake and appetite. Physiol Behav. 2021 Dec 1;242:113622. doi: 10.1016/j.physbeh.2021.113622. Epub 2021 Oct 12. PMID 34653498
- See also: Full4Health web-site — http://www.full4health.eu/